CLINICAL TRIAL: NCT06181071
Title: Investigation of the Acute Effects of Distal and Proximal Muscle Fatigue on the Mechanical and Viscoelastic Properties of Lower Extremity, Foot Pressure Distribution, and Balance in Healthy Young Adults
Brief Title: Effectiveness of Distal and Proximal Muscle Fatigue for Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gülenay Yıldırım, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SaglikBilimleri22-114
Record Dates: First submitted 2023-12-11; First posted 2023-12-26 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Young Adult; Fatigue
Keywords: muscular fatigue; balance; elasticity; muscle tonus; foot plantar pressure
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Distal Fatigue of The Lower Extremity (Other): Distal muscle fatigue of the lower extremity involves the plantar and dorsiflexor muscles of the ankle.
  Interventions: Other: Distal Muscle Fatigue Protocol; Other: Proximal Muscle Fatigue Protocol
- Proximal Fatigue of The Lower Extremity (Other): Proximal muscle fatigue of the lower extremity involves hip flexor and extansor muscles.
  Interventions: Other: Distal Muscle Fatigue Protocol; Other: Proximal Muscle Fatigue Protocol

INTERVENTIONS:
Other: Distal Muscle Fatigue Protocol — Initially, sociodemographic data, muscle viscoelastic properties, foot plantar pressure, and static and dynamic balance are assessed. Additionally, the strengths of the plantar flexor and dorsiflexor muscles are evaluated. After these assessments, the heel raise exercise will be implemented in this protocol. Firstly, dominant leg, the heel raise exercise will be performed for 3 sets with the knees in full extension until the individual reaches fatigue. Subsequently, the heel raise exercise will be conducted for another 3 sets with the knee in flexion until the individual reaches fatigue. Following these exercises, Then, the strengths of the hip flexor and extensor muscles will be re-evaluated. If the individual reports a value of 7 or higher on the modified Borg scale, the viscoelastic properties of the muscles, foot plantar pressure, and static and dynamic balance will be reassessed when a 50% decrease in the initial strength is detected.
Other: Proximal Muscle Fatigue Protocol — One week after the application of the distal muscle fatigue protocol, the same individuals will undergo the proximal fatigue protocol. In this protocol, individuals will perform, dominant leg, a single-leg squat exercise targeting the fatigue of the hip flexor and extensor muscles. Prior to this exercise, the viscoelastic properties of the muscles, foot plantar pressure, static and dynamic balances, as well as the strengths of the hip flexor and extensor muscles will be assessed. Then, individuals will perform the single-leg squat exercise, 3 sets. When the individual indicates fatigue, the set will conclude, allowing a 30-second rest between sets. Then, the strengths of the hip flexor and extensor muscles will be re-evaluated. If the individual reports a value of 7 or higher on the modified Borg scale, the viscoelastic properties of the muscles, foot plantar pressure, and static and dynamic balance will be reassessed when a 50% decrease in the initial strength is detected.

SUMMARY:
This is a study aiming to investigate the effects of acute muscle fatigue on muscle properties, balance and foot plantar pressure in healthy young adults (having no chronic diseases or orthopaedic diseases and physically active). This study also aims to compare the effects of foot muscle fatigue and hip muscle fatigue on balance and foot plantar pressure.

The exercises for ankle muscle fatigue are heel rise with bending your knee and heel raise without bending your knees.

The exercise for hip muscle fatigue is a single-leg squat. Before and after completing these all exercises, the balance is evaluated with an isokinetic balance device, the foot plantar pressure is evaluated with a pedobarography device and finally, the muscle properties are evaluated with a myotonPro device. All assessment devices are non-invasive.

DETAILED DESCRIPTION:
The International Physical Activity Questionnaire (Short form) will be used to assess individuals' physical activity levels. Prior to the distal and proximal fatigue protocols, the participants' maximum isometric muscle forces of the gastrocnemius, soleus, tibialis anterior, rectus femoris, and gluteus maximus muscles will be evaluated using a dynamometer.

Then, the mechanical and viscoelastic properties of these muscles and the iliotibial band will be assessed using the MyotonPro device, participants' static foot pressure on both feet will be evaluated through pedobarography, and individuals' dynamic balance and static balance will be evaluated on one foot using the Technobody isokinetic balance device.

The individuals included in the study will undergo exercises targeting the foot plantar flexor and dorsiflexor muscles on the first day, and exercises targeting the hip flexor and extensor muscles on the second day. The researcher will measure the voluntary maximum isometric muscle strength using a dynamometer,

Heel raise exercises will be performed in 3 sets, with 30 seconds of free walking allowed for rest between sets. Individuals will initially complete 3 sets of this exercise without bending their knees. Then, they will perform the heel raise exercise with bent knees. The researcher will measure the voluntary maximum isometric muscle strength using a dynamometer when the Modified Borg Scale indicates a level of 7 or above. If the muscle strength has decreased to 50% of the initial force, indicating fatigue, the exercise will be terminated.

Second day, a single-leg squat will be performed in 3 sets, with 30 seconds of free walking allowed for rest between sets.The researcher will measure the voluntary maximum isometric muscle strength using a dynamometer when the Modified Borg Scale indicates a level of 7 or above. If the muscle strength has decreased to 50% of the initial force, indicating fatigue, the exercise will be terminated.

After the distal fatigue protocol, the viscoelastic properties of the gastrocnemius, soleus, and tibialis anterior muscles will be assessed using the MyotonPro device, while the plantar pressures will be evaluated through pedobarography. Additionally, static and dynamic balances will be measured using the Technobody device. Following the proximal fatigue protocol, the mechanical and viscoelastic properties of the gluteus maximus and rectus femoris muscles, along with the iliotibial band, will be examined using the MyotonPro device. Similarly, plantar pressures will be analyzed through pedobarography, and static and dynamic balances will be assessed using the Technobody device. The collected data will be recorded by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* To be a healthy individual in the age range of 18-35,
* To be willing to participate in the study,
* To have a minimal active or highly active score on the International Physical Activity Questionnaire (Short Form),
* To have a body mass index (BMI) of 24.9 kg/m² or lower.

Exclusion Criteria:

* Having a history of injury and/or surgical operation related to the lower extremity,
* Having limited mobility in the lower extremity,
* Having any deformity related to the lower extremity,
* Having cardiovascular, vestibular, neurological, orthopedic, or skin-related diseases,
* Having any chronic disease that may affect balance,
* Having any acute/chronic musculoskeletal pain or systemic pain,
* Not to have given consent to participate in the study or to wish to withdraw from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Myotonometric Assesment | Day 1 and Day 8
  Myotonometeric assessment is a non-invasive and novel method used to characterize the viscoelastic and biomechanical properties of muscles. The MyotonPro (Myoton Ltd, Myoton AS, Estonia) is an objective assessment tool that has been validated for inter-rater and intra-rater reliability, enabling the evaluation of mechanical and viscoelastic properties such as muscle tone, stiffness, and elasticity. The MyotonPro device is positioned perpendicular to the skin surface when the muscles are in a relaxed position. The device's probe applies an initial pressure of approximately 0.18 N to the skin surface, compressing the underlying tissue. Subsequently, a mechanical force of 0.4 N is applied for 15 ms to the compressed tissue beneath the skin.
Isokinetic Balance Assesment | Day 1 and Day 8
  The TecnoBody Prokin PK 252 device, which is one of the objective methods used for the assessment of static and dynamic balance, allows the acquisition of numerical data at the end of the evaluation. Equipped with an isokinetic balance system, this device consists of a screen monitor and a sloped platform on which the individuals being evaluated stand. This platform has air pistons that provide a 15-degree tilt in all directions. These air pistons come into play, especially during the assessment of dynamic balance. The settings of the platform can be adjusted according to the evaluator's decision, thanks to the servo motors associated with the device.

SECONDARY OUTCOMES:
Foot Plantar Pressure Distribution Assesment | Day 1 and Day 8
  The analysis of foot plantar pressure distrubition is conducted using the objective and valid method of pedobarography. The Sensor Medica device, specifically the FreeStep v.1.0.3 88 software (Sensor Medica, Guidonia Montecelio, Rome, Italy), has been utilized for the analysis of pressure distributions. This device features a FreeMed Maxi Baropodometric Platform made of aluminum. The FreeStep software is employed for pressure analysis. Through this platform and the FreeStep software, foot plantar pressure distrubition can be assessed both statically and dynamically.

CONTACTS AND LOCATIONS:
Overall Officials: Gulenay Yildirim, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation Laboratory, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No